CLINICAL TRIAL: NCT00116246
Title: McRoberts Manoeuvre Or Pushing Study (McMOPS)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Melbourne (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 02151B
Record Dates: First submitted 2005-06-27; First posted 2005-06-28 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2005-08

CONDITIONS: Childbirth
Keywords: Labour; vaginal delivery; primigravida; McRobert's Manoeuvre; operative delivery

INTERVENTIONS:
Procedure: McRobert's manoeuvre

SUMMARY:
We propose to conduct a randomised-controlled study to investigate whether adopting McRoberts' position, after 45 minutes of active pushing with no signs of progress, can increase the probability of vaginal delivery, preventing the need for forceps or vacuum assistance. In our study we will allow 45 minutes of pushing before a further 45 minutes of either the same, or our intervention (McRoberts' manoeuvre).

DETAILED DESCRIPTION:
When women are in labour, they firstly undergo the first stage of labour where the cervix (neck of the womb) progresses to full dilatation. Once this occurs, they have reached the second stage, where the mother can start pushing to deliver the baby. It is accepted practice to allow mothers to actively push for a maximum of one hour.

In most cases, the baby will deliver spontaneously. However, in about 30% of cases of those who manage to labour to the second stage (fully dilated cervix), the obstetrician will have to assist delivery by the use of forceps or vacuum extraction (instrumental delivery). There are two main situations where delivery needs assistance; 'fetal distress' where the baby is suspected to be compromised, or failure to progress where the baby has not delivered after one hour of pushing. Unfortunately, instrumental delivery is associated with increased maternal and fetal problems, particularly arising from trauma to the tissues. Therefore, the identification of any new ways to increase the spontaneous delivery rate may decrease future complications.

Shoulder dystocia is a rare but dangerous scenario where the baby's head is delivered, but the shoulders are trapped behind the pubic bones. The McRoberts' position is used in this situation to deliver the baby. The mother's legs are flexed, and pushed up and out, lateral to her abdomen. It is believed that this helps by flattening out the sacral bone (tail bone), thereby widening the bony opening and allowing the shoulders to become free.

A recent paper (1) reported the novel finding that McRoberts' position also doubled the pressure generated by contractions compared to normal pushing. The authors believed that this increase in pressure was caused by the fact that the uterus was brought closer to the diaphragm that provides the power generated with pushing.

Our group wondered whether this substantial increase in pressure could be harnessed beyond the rare setting of shoulder dystocia. We therefore propose to conduct a randomised-controlled study to investigate whether adopting McRoberts' position, after 45 minutes of active pushing with no signs of progress, can increase the probability of vaginal delivery, preventing the need for forceps or vacuum assistance. Studies have shown that after one hour of active pushing, the fetus shows signs of increasing distress. In our study we will allow 45 minutes of pushing before a further 45 minutes of either the same, or our intervention (McRoberts' manoeuvre).

Women in their first pregnancy will be approached at 36 weeks in the antenatal clinic and advised of our study in the form of written information. The majority of women will not be approached again since they will not be relevant to this study, most having already delivered. However, women who have been pushing for 45 minutes will be invited to participate in the study.

The second stage of labour is a demanding process where it may not be practicable to obtain written consent. Therefore, having given information about the trial at their 36 week antenatal visit, we will enrol women after obtaining informed verbal consent. They will be specifically asked whether they have read and understood the prior information given to them at clinic.

Those consenting will be randomised to either continue in their current position or be placed in McRoberts' position. The woman will be allowed to push for a further 45 minutes. After this time, women in both groups who have not yet delivered will be aided by instrumental delivery, if deemed necessary. A few days after delivery, we will provide women with a questionnaire to determine patient satisfaction and how well they tolerated the procedure they ended up having (i.e. Operative delivery or McRoberts position).

We hope to find a significant reduction in the number of instrumental deliveries in the group of women placed in McRoberts' position as compared with the other group. A positive finding may be immediately, and widely applicable.

References:

1. Catalin, SB et al, "Use of McRoberts' position during delivery and increase in pushing efficiency", The Lancet (2001); 358: 470-471
2. Nordstrom L et al, "Fetal and maternal lactate increase during active second stage of labour", British Journal of Obstetrics and Gynaecology, (2001); 108;263-268.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women in labour after 37 completed weeks gestation who have been pushing for 45 minutes in the second stage of labour with no progress (defined as no presenting part visible on pushing, without parting the labia)
* Singleton pregnancy
* Cephalic presentation
* Clinical scenarios in which we propose to still include in the study: *Spontaneous or induced labour; *Regional anaesthesia; *Clinical suspicion of large baby, but was considered suitable for trial of labour

Exclusion Criteria:

* Maternal weight >100kgs
* Non-reassuring fetal condition
* Patient being unable to tolerate McRobert's position
* Non-English speaking woman
* Woman unable to give adequate consent, or suspicion that the antenatal information sheet has not been fully understood
* Multiparous women
* Complicated obstetric co-morbidities, including: *Preterm labour (less than 37 completed weeks gestation); *Multiple pregnancy; *Abnormal presentation; *Placenta praevia or abruption; *Non-reassuring fetal status Maternal pathology restricting maternal adoption of McRoberts' position (e.g. back problems)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 222
Dates: Start 2005-08; Study Completion 2006-12

PRIMARY OUTCOMES:
Operative delivery rate
Patient satisfaction with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sheila F Mulvey, PhD,MB, Principal Investigator — University of Melbourne,Dept of Obstetrics & Gynaecology
Locations (1):
- Mercy Hospital for Women, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Buhimschi CS, Buhimschi IA, Malinow A, Weiner CP. Use of McRoberts' position during delivery and increase in pushing efficiency. Lancet. 2001 Aug 11;358(9280):470-1. doi: 10.1016/S0140-6736(01)05632-X. PMID 11513914
- [Background] Murphy DJ. Failure to progress in the second stage of labour. Curr Opin Obstet Gynecol. 2001 Dec;13(6):557-61. doi: 10.1097/00001703-200112000-00002. PMID 11707657
- [Background] Nordstrom L, Achanna S, Naka K, Arulkumaran S. Fetal and maternal lactate increase during active second stage of labour. BJOG. 2001 Mar;108(3):263-8. doi: 10.1111/j.1471-0528.2001.00034.x. PMID 11281466
- [Background] Robinson JN, Norwitz ER, Cohen AP, McElrath TF, Lieberman ES. Episiotomy, operative vaginal delivery, and significant perinatal trauma in nulliparous women. Am J Obstet Gynecol. 1999 Nov;181(5 Pt 1):1180-4. doi: 10.1016/s0002-9378(99)70104-3. PMID 10561641